CLINICAL TRIAL: NCT04049851
Title: Randomized Clinical Trial, Double-blind, Single-dose Drug and Escalating Infection Intensities, Evaluating the Safety and Efficacy of Moxidectin 2 mg, Ivermectin-controlled, in Loa Loa Microfilaremic Patients
Brief Title: Clinical Trial Evaluating the Safety and Efficacy of Moxidectin 2 mg Ivermectin-controlled in Loa Loa Microfilaremic Patients
Acronym: EOLoa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center for Research on Filariasis and Other Tropical Diseases, Cameroon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C18-57
Record Dates: First submitted 2019-07-26; First posted 2019-08-08 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Onchocerciasis, Ocular; Loiasis
MeSH Terms: conditions — Onchocerciasis, Ocular; Loiasis | interventions — moxidectin; Tablets; Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moxidectin (Experimental)
  Interventions: Drug: Moxidectin 2 MG Oral Tablet; Drug: Placebo oral tablet
- Ivermectin (Active Comparator)
  Interventions: Drug: Ivermectin 3Mg Tab; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Moxidectin 2 MG Oral Tablet — One Moxidectin 2 mg tablet will be blinded and will be administrated with 3 tablets of placebo.
  Arms: Moxidectin
Drug: Ivermectin 3Mg Tab — 3 ivermectin tablets (or 4 according to the weight) will be blinded and will be administrated with 1 (or 0 according to the weight) tablet of placebo.
  Arms: Ivermectin
Drug: Placebo oral tablet — Placebo will be administrated with Moxidectin or ivermectin. Each participant will have 4 tablets in total.

SUMMARY:
This study aims at evaluating the safety and efficacy of Moxidectin 2 mg in patients with low intensities of microfilariae of Loa loa.

DETAILED DESCRIPTION:
This clinical trial will be randomized, double blind, and will compare Moxidectin to ivermectin. This study will be conducted in Cameroon.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent written, signed (or with a cross) and dated
* Men aged 18 to 65 included (women not included in the study)
* Microfilarial density between 1 and 1,000 mf/mL
* body weight ≥ 45 kg and less than 85 kg
* Good general condition, as determined by the medical questionnaire and clinical examination
* Hematological parameters and adequate renal and hepatic functions, such as:

  * Leukocytes ≥ 2,800 and ≤ 11,300 cells/mL
  * Hemoglobin ≥ 10.0 g/dL
  * Platelets ≥100,000/mm3
  * Serum creatinine ≤ 2.5 upper limit (UL) of the laboratory
  * Total bilirubinemia ≤ 2.5 x UL
  * ALAT ≤ 2.5 x UL
  * Negative urinary strip: absence of leucocyturia, hematuria, and proteinuria (in case of positivity, a second urinary strip test will be made, for confirmation)

Exclusion Criteria:

* Participation in any study other than purely observational, in the 4 weeks preceding this study (determined by the theoretical date of administration of MOX-2 mg or IVM).
* Person who has taken IVM in the last 6 months
* Any vaccination in the 4 weeks preceding this study
* Acute infection requiring a treatment in the 10 days preceding this study, determined by the anamnesis during the medical interview (example: pulmonary infection, ENT, digestive, cutaneous, with implementation of an antibiotic treatment or not)
* Long-term antiretroviral therapy (protease inhibitor, non-nucleoside reverse transcriptase inhibitor), or treatment with ampicillin or chloramphenicol within 10 days prior to administration of the test drug
* History or presence of neurological (including epilepsy) or neuropsychiatric disease
* Excessive consumption of alcohol or other drug abuse within 72 hours prior to the administration of the test treatment determined by the medical history during the medical interview.
* Any condition, in the opinion of the investigator, which exposes the subject to an undue risk
* Subjects who donated blood in the 8 weeks prior to study entry, with a standard volume (> 500 mL)
* Known intolerance to IVM, MOX or any of the excipients (including placebo)
* During the clinical examination: symptoms, physical signs or biological constants suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, cutaneous, immunodeficiency, psychiatric disorders and other abnormalities likely to interfere with the interpretation results of the test. The doctor may then give a favorable or unfavorable opinion for the inclusion of the participant

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Incidence of severe adverse events post Moxidectin 2 mg | 1 week
  Absence of severe adverse events
Incidence of adverse events with Moxidectin 2 mg | 1 week
  Proportion of adverse events during the first week

SECONDARY OUTCOMES:
Proportion of reduction of the microfilarial densities of Loa loa : short term efficacy | Day 7 and Day 15
  Proportion of reduction of the microfilarial densities of Loa loa at Day 7 and Day 15
Proportion of reduction of the microfilarial densities of Loa loa : long term efficacy | Day 80, Day 180, and Year 1
  Proportion of reduction of the microfilarial densities of Loa loa at Day 80, Day 180, and Day 365
Percentage of individuals without microfilaria post Moxidectin 2 mg | Day 7, Day 90, Day 180, and Year 1
  Percentage of individuals without microfilariae of Loa loa at Day 7, Day 90, Day 180, and Day 365

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche sur les filarioses et autres maladies tropicales (CRFilMT), Yaoundé, Cameroon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wafeu GS, Lepage TM, Campillo JT, Efon-Ekangouo A, Nana-Djeunga HC, Nzune-Toche N, Domche A, Sumo L, Njitchouang GR, Tsasse MAF, Bopda J, Balog YA, Niamsi-Emalio Y, Mbickmen-Tchana S, Talla GK, Kana YSN, Messina FDM, Pion SD, Kuesel AC, Kamgno J, Boussinesq M, Chesnais CB. Safety and Short-term Efficacy of a Single Dose of 2 mg Moxidectin in Loa loa-Infected Individuals: A Double-Blind, Randomized Ivermectin-Controlled Trial With Ascending Microfilarial Densities. Open Forum Infect Dis. 2024 Apr 25;11(7):ofae240. doi: 10.1093/ofid/ofae240. eCollection 2024 Jul. PMID 38966851